CLINICAL TRIAL: NCT02574689
Title: Home-based, Individually-tailored Physical Activity Print Intervention for African American Women in the Deep South
Acronym: HIPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Dorothy Pekmezi, PhD, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: X130405004
Record Dates: First submitted 2015-09-15; First posted 2015-10-14 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Physical Activity
Keywords: Physical Activity; Cancer Prevention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIPP Intervention (Experimental): The physical activity intervention emphasizes behavioral strategies for increasing activity levels (i.e., goal-setting, self-monitoring, problem-solving barriers, increasing social support, rewarding oneself for meeting physical activity goals), and includes regular mailings (three mailings in month 1, two mailings in months 2 and 3, one mailing in months 4, 5, 6, 8, and 10) of physical activity manuals that are matched to the participant's current level of motivational readiness and individually-tailored computer expert system feedback reports.
  Interventions: Behavioral: HIPP
- Wellness Contact Control (Active Comparator): Cancer prevention information on topics other than physical activity (e.g., "Add Fruits and Veggies to Your Diet") from the ACS website (www.cancer.org) will be mailed to control participants at the same time points that the HIPP Intervention participants receive their physical activity intervention materials.
  Interventions: Behavioral: Wellness contact control

INTERVENTIONS:
Behavioral: HIPP — The physical activity intervention is based on the Social Cognitive Theory and Transtheoretical Model and includes motivation-matched physical activity manuals and individually-tailored computer expert system feedback reports. Tailored reports are based on participants' monthly update survey data and cover: 1) current stage of change; 2) self-efficacy; 3) decisional balance; 4) social support; 5) outcome expectations; 6) enjoyment; 7) progress feedback; 8) normative feedback; 9) self regulation. The computer expert system draws from a bank of 330 messages addressing different levels of psychosocial and environmental factors affecting physical activity.
  Arms: HIPP Intervention
Behavioral: Wellness contact control — Cancer prevention information on topics other than physical activity (e.g., "Add Fruits and Veggies to Your Diet") from the American Cancer Society website (www.cancer.org) are mailed to control participants at the same time points that the HIPP Intervention participants receive their physical activity intervention materials.
  Arms: Wellness Contact Control

SUMMARY:
This pilot study represents an initial foray into delivering home-based individually-tailored physical activity interventions for cancer risk reduction among African American women in the Deep South.

DETAILED DESCRIPTION:
80 women will receive the HIPP Intervention or Wellness Contact Control. While main outcomes are focused on feasibility and acceptability, physical activity, fitness, and body weight and composition data will be collected at baseline, 6 months, and 12 months, along with blood draws.

HIPP Intervention: The physical activity intervention is based on the Social Cognitive Theory and Transtheoretical Model and, emphasizes behavioral strategies for increasing activity levels (i.e., goal-setting, self-monitoring, problem-solving barriers, increasing social support, rewarding oneself for meeting physical activity goals), and includes regular mailings (three mailings in month 1, two mailings in months 2 and 3, one mailing in months 4, 5, 6, 8, and 10) of physical activity manuals that are matched to the participant's current level of motivational readiness and individually-tailored computer expert system feedback reports. Computer expert system feedback reports will be based on participants' monthly update survey data and include information on:

1. current stage of motivational readiness for physical activity;
2. increasing self- efficacy (i.e., confidence) for physical activity participation;
3. weighing the pros and cons of engaging in physical activity (decisional balance);
4. social support from family and friends for physical activity participation;
5. outcome expectations (beliefs regarding the consequences of physical activity participation);
6. perceived enjoyment of physical activity;
7. how the participant compares to her prior responses (progress feedback);
8. how the participant compares to individuals who are physically active and with national guidelines (normative feedback);
9. self monitoring of physical activity behavior (using pedometers and activity logs to track the total steps and minutes of moderate intensity physical activity per day).

The computer expert system draws from a bank of 330 messages addressing different levels of psychosocial and environmental factors affecting physical activity. Intervention participants will also receive tip sheets addressing physical activity barriers specific to African American women in the Deep South (as identified during our focus groups and comprehensive literature review).

Wellness Contact Control Condition: Cancer prevention information on topics other than physical activity (e.g., "Add Fruits and Veggies to Your Diet") from the American Cancer Society (ACS) website (www.cancer.org) will be mailed to control participants at the same time points that the HIPP Intervention participants receive their physical activity intervention materials.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Post-menopausal (defined as not having menstrual periods for at least 12 months)
* Not taking hormone replacement therapy
* Healthy (BMI 18.5-40; No history of heart disease, myocardial infarction, angina, stroke, or orthopedic conditions which limit mobility, or any serious medical condition that would make physical activity unsafe; no psychiatric hospitalization in past 3 years).
* Not taking medication that may impair physical activity tolerance or performance (e.g., beta blockers).
* Not planning to move from the area for the next 12 months
* Willing to be randomized to either study arm and adhere to study protocol

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2014-09; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
7-Day Physical activity Recall interview (change from baseline in 7-Day physical activity recall interview) | baseline and 6 months
  minutes/week of moderate intensity or greater physical activity
7-Day Physical activity Recall interview (change from baseline in 7-Day physical activity recall interview) | baseline and 12 months
  minutes/week of moderate intensity or greater physical activity

SECONDARY OUTCOMES:
6 minute walk test | baseline, 6 months, 12 months
  meters walked in 6 minutes
body mass index | baseline, 6 months, 12 months
  kg/m^2
waist circumference | baseline, 6 months, 12 months
  cm
body impedance analyses | baseline, 6 months, 12 months
  % body fat
Social Support for exercise scale | baseline, 6 months, 12 months
  range=0-65 for both friends and family subscales, with higher scores indicating more social support
Outcome expectations scale | baseline, 6 months, 12 months
  range= 1-5, with higher scores representing more outcome expectations
Physical Activity Enjoyment scale | baseline, 6 months, 12 months
  range=18-126, with higher scores indicating more enjoyment
accelerometers | baseline, 6 months, 12 months
  minutes/week of moderate intensity or greater physical activity
Stages of Readiness Measure | baseline, 6 months, 12 months
  categorize participants into stages of change (pre contemplation, contemplation, preparation, action, maintenance)
Self -Efficacy for physical activity scale | baseline, 6 months, 12 months
  range= 1-5, with higher scores representing more self-efficacy
processes of change measure | baseline, 6 months, 12 months
  range= 1-5, with higher scores representing greater use of cognitive and/or behavioral processes of change
Decisional Balance scale | baseline, 6 months, 12 months
  scores >0 indicate more advantages than disadvantages to physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Dori Pekmezi, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States